## WAIVER OF DOCUMENTATION OF CONSENT

INVESTIGATOR'S NAME: DEBRA PARKER OLIVER, PHD

PROJECT # 2003012

## STUDY TITLE: SHARED DECISION MAKING TO IMPROVE PALLIATIVE CARE IN THE NURSING HOME

- 1. I would like to ask you to participate in a study that involves research.
- 2. Participation is voluntary and your decision not to participate will not involve any penalty or loss of benefits *and will in no way affect the nursing home care you receive*.
- 3. For this study, your family member will be asked to answer questions about their experience with you in the nursing home.
- 4. The purpose of our study is to investigate ways to improve nursing home care by including residents and family in the care plan meeting.
- 5. We are asking approximately 46 residents and their family to participate in this study.
- 6. The study staff may withdraw you from the study at any time after explaining to you the reason for withdrawal.
- 7. While on the study, you are at risk for some people may experience frustration using technology with which they may not be familiar or may feel anxious or uneasy participating in team meetings. Please do not hesitate to discuss your concerns or concerns related to the questions with the research staff.
- 8. If you agree to take part in this study, there may or may not be direct medical benefit to you. If you are assigned to the intervention group, you will have access to the nursing home team and your family member. We hope the information learned from this study will benefit other nursing home residents and their family.
- 9. If you choose to participate, Information produced by this study will be stored in the investigator's locked file or secured computer and identified by a code number only. The code key connecting your name to specific information about you will be kept in a separate, secure location. Information contained in your records may not be given to anyone unaffiliated with the study in a form that could identify you without your written consent, except as required by law. All research materials, including the video recordings and transcripts will be maintained for 7 years following the completion of the study. The results of this study may be published in a medical book or journal or used for teaching purposes. However, your name or other identifying information will not be used in any publication or teaching materials without your specific permission.
- 10. There is no cost to you for the participating in the study. However, you will still be paying for the normal cost of your routine nursing home.

MU: Waiver of Documentation of Consent

IRB USE ONLY

Approval Date: December 12, 2016

**Expiration Date: November 20, 2017** 

- 10. There is no compensation given to you for participation in this study, however your family will receive \$50 for their participation.
- 11. If you have any questions regarding your rights as a participant in this research and/or concerns about the study, or if you feel under any pressure to enroll or to continue to participate in this study, you may contact the University of Missouri Health Sciences Institutional Review Board (which is a group of people who review the research studies to protect participants' rights) at (573) 882-3181.
- 12. If you have any problems or questions, you may contact Debra Parker Oliver 573-884-53011 would be happy to answer any questions that you may have.
- 13. A copy of this script will be given to you to keep

MU: Waiver of Documentation of Consent

IRB USE ONLY

Approval Date: December 12, 2016 Expiration Date: November 20, 2017